CLINICAL TRIAL: NCT04692896
Title: Effect of Different Concentrations of Lidocaine in Relieving Pain Peroperatively and 24 Hours Postoperatively in Wide Awake Hand Surgery Using Tumescent Local Anesthesia Technique
Brief Title: Effect of Different Concentrations of Lidocaine in Relieving Pain in Wide Awake Hand Surgery Using Tumescence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mustehsan Bashir, Professor of Plastic Surgery, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 27/RC/KEMU
Record Dates: First submitted 2020-12-27; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Lidocaine
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 0.1% lidocaine (Experimental)
  Interventions: Drug: lidocaine
- 0.2% lidocaine (Experimental)
  Interventions: Drug: lidocaine
- 0.3% lidocaine (Experimental)
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — different concentrations of lidocaine with same concentration of adrenaline
  Other Names: adrenaline

SUMMARY:
Lidocaine has been used along with adrenaline in tumescent anesthesia for a variety of procedures. This has been quite popular especially in wide awake surgery of the hand with no tourniquet. However, the appropriate lidocaine concentration is yet to be established. This randomized control trial will study the minimum effective lidocaine concentration in hand surgery using the tumescent technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 16 to 60 years of either gender
2. Patients with post burn/post traumatic contractures involving fingers & palm
3. Patients with nerve injury or flexor/extensor tendons injury distal to mid forearm.

Exclusion Criteria:

1. Patients with history of ischemic heart disease, chronic liver disease (ALT/AST 40 IU/L), renal disease (creatinine 13mg/dl), bleeding disorder, peripheral arterial disease & peripheral neuro3pathy .
2. Surgical site infection .
3. History of allergic hypersensitivity to epinephrine or lidocaine.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
total duration of analgesia | Within 24 hours of randomization.
  Patients were randomized to either 0.1percent, 0.2 percent and 0.3 percent groups. Tumescent local anesthesia was infiltered. Surgery was started approximately 25 minutes after the infiltration. Start of surgery was designated 0 minute. Duration of pain free surgery was noted in minutes. Pain scores was measured after surgery. When pain scores was equal to or more than 4, analgesia was given and total time in minute from start of surgery till this time was taken as total duration of analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of plastic Surgery,Mayo Hospital King Edward Medical University, Lahore, Pujab, Pakistan